CLINICAL TRIAL: NCT05499546
Title: Polyp Size Measurement During Real-time Colonoscopy Using the Virtual Scale Function SCALE EYE: Variability and Systematic Differences
Brief Title: Virtual Scale Function SCALE EYE: Variability and Systematic Differences
Acronym: SCALE-EYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL81269.018.22
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Polyp of Colon
Keywords: Colorectal polyp; Size; SCALE EYE; Virtual scale
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): All patients within the study are included in the intervention arm: polyp detected within these patients will be measured according to the study protocol using four different methods.
  Interventions: Device: SCALE EYE

INTERVENTIONS:
Device: SCALE EYE — Polyp size measurement using the SCALE EYE functionality

SUMMARY:
Size of colorectal polyps is important to decide on appropriate surveillance intervals and treatment modality, as well as carrying out optical diagnosis strategies. However, polyp size measurement is often prone to inter-observer variability. An easy and accurate tool to assist in polyp size measurement is required. Recently, a virtual scale function for size measurement during endoscopy (SCALE EYE), operating in real-time without the use of any additional devices, has been developed. The aim of this study is to assess whether use of the SCALE EYE for polyp size measurement can reduce inter-observer variability.

DETAILED DESCRIPTION:
This study is designed as a single center prospective study. Polyp size measurements using SCALE EYE will be compared with several other polyp size measurement techniques: size measurements by endoscopists without a reference ('carpenters eye') , size measurements by endoscopists with an opened snare (of known size) as reference and size measurements by the pathologist during histopathological analysis.

During screening colonoscopies, detected polyps (maximum of four per colonoscopy) will be measured using all three different colonoscopy measurement techniques. This will be done by experienced endoscopists (endoscopist accredited for colonoscopies within the national colorectal cancer screening program). Since endoscopists measure polyps in multiple ways, consecutive measurements of the same polyp will be biased. For this reason, all polyp size measurements will be recorded on video. The video recordings of the different measurements of all polyps will be presented to eight expert endoscopists and four to eight trainees (depending on availability) in a randomized order. The size estimations based on these video recordings will be used for further analysis. Histopathological analysis and size measurements of the resected polyps will be performed by pathologists with expertise in gastrointestinal pathology. Variability and systematic differences in polyp size measurement between different measurements methods will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Screening colonoscopy after positive fecal immunochemical test (FIT) within the Dutch colorectal cancer screening program
* Signed informed consent

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease, Lynch syndrome or (serrated) polyposis syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Differences in residual variance expert endoscopists | Through study completion, an average of 3 months
  The difference in residual variance (variability) between (1) polyp size measurement with SCALE EYE and (2) polyp size measurement using an opened snare (of known size) as reference.

SECONDARY OUTCOMES:
Differences in residual variance expert endoscopists | Through study completion, estimation: 3 months
  The difference in residual variance (variability) between polyp size measurement with (1) the SCALE EYE functionality, (2) polyp size measurement without reference and (3) polyp size measurement during histopathological analysis.
Systematic differences expert endoscopists | Through study completion, estimation: 3 months
  The systematic difference in polyp size measurements between (1) the SCALE EYE functionality and the other measurement techniques: (2) polyp size measurement without reference, (3) polyp size measurement with an opened snare as a visual reference and (4) polyp size measurement during histopathological analysis.
Differences in residual variance and systematic differences trainees | Through study completion, estimation: 3 months
  Aforementioned parameters / outcomes (and primary study parameter) based on assessment by trainees (for other analyses assessment by experts will be used).
Inter-observer variability | Through study completion, estimation: 3 months
  Inter-observer variability within techniques (residual variance).
SCALE EYE measurement accuracy compared to snare measurement | Through study completion, estimation: 3 months
  The accuracy of the SCALE EYE functionality for predicting the size of polyps. Accuracy is defined as the percentage of correctly predicted polyp sizes with the SCALE EYE functionality when polyp size measurement with an opened snare is considered as reference standard. Polyp size will be assigned as correctly predicted if the polyp size measurement with SCALE EYE lies within a 25% margin of error. The mean of the polyp size measurements by all experts endoscopists will be used for the comparison.
SCALE EYE measurement accuracy compared to snare measurement for different polyp size groups | Through study completion, estimation: 3 months
  The accuracy of the SCALE EYE functionality for predicting polyp size for different polyp size categories (1-5 mm vs. 6-9 mm vs. >10 mm). Accuracy is defined as the percentage of correctly predicted polyp sizes with the SCALE EYE functionality when polyp size measurement with an opened snare is considered the reference standard. Polyp size will be assigned as correctly predicted if the polyp size measurement with SCALE EYE lies within a 25% margin of error. The mean of the polyp size measurements by all expert endoscopists will be used to assign the polyp size category.
SCALE EYE success rate | Through study completion, estimation: 3 months
  The proportion of successful polyp size measurements by SCALE EYE during live endoscopy.
SCALE EYE measurement time | Through study completion, estimation: 3 months
  Average time to manoeuver SCALE EYE during live endoscopy (i.e. time to perform measurement of one polyp).
SCALE EYE satisfaction score | Through study completion, estimation: 3 months
  Satisfaction score for usage of SCALE EYE (scale from 1-10).

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Dekker, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Bergman Clinics, Amsterdam, Norod-Holland
  - Academic Medical Centre, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Bokhorst QNE, Houwen BBSL, Hazewinkel Y, van der Vlugt M, Beaumont H, Grootjans J, van Tilburg A, Fockens P, Bossuyt PMM, Dekker E; SCALE EYE study group. Polyp size measurement during colonoscopy using a virtual scale: variability and systematic differences. Endoscopy. 2025 Feb;57(2):137-145. doi: 10.1055/a-2371-3693. Epub 2024 Jul 23. PMID 39043201